CLINICAL TRIAL: NCT07260825
Title: Use of Topical Testosterone and Estrogen vs Estrogen Alone in Vulvodynia: a Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-108
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Vulvodynia; Dyspareunia; Lichen Sclerosus of Vulva
Keywords: topical testosterone; estrogen cream; vulvodynia
MeSH Terms: conditions — Vulvodynia; Dyspareunia; Vulvar Lichen Sclerosus | interventions — Estradiol; Vaginal Creams, Foams, and Jellies; Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (Active Comparator): Patients receiving standard of care
  Interventions: Drug: Estradiol 0.01% Vag Cream
- Treatment (Experimental): Patients receiving study treatment
  Interventions: Drug: testosterone 0.1% and estradiol 0.01% vaginal cream

INTERVENTIONS:
Drug: Estradiol 0.01% Vag Cream — 0.01% Estradiol cream, 1g to be applied to the vestibule twice daily for 12 weeks
  Arms: Standard of care
Drug: testosterone 0.1% and estradiol 0.01% vaginal cream — 0.01% Estradiol and 0.1% testosterone cream, apply 1g to the vestibule twice daily for 12 weeks
  Arms: Treatment

SUMMARY:
We are looking to see if patients using both topical testosterone and estrogen will have a greater improvement in pain with vaginal penetration compared to those using topical estrogen alone.

DETAILED DESCRIPTION:
You are being asked to take part in this research study because you have vulvodynia. Vulvodynia refers to pain in the female vestibule. The vestibule is the area that encircles the vaginal opening and the urethra opening. One of the symptoms of vulvodynia is pain with intercourse.

The purpose of this research study is to determine if using estrogen cream versus a combined cream with estrogen and testosterone helps decrease your pain with intercourse.

Multiple studies have been conducted looking at the use of combined cream with estrogen and testosterone to treat vulvodynia. However, none of the studies have compared this to using estrogen cream alone. It is well known that estrogen cream applied to the vagina helps reduce symptoms of vulvodynia. Combined creams with estrogen and testosterone have been shown to help patients who have vulvodynia and are taking birth control pills.

In 2016, the FDA approved a vaginal cream, known as DHEA, to help women with painful intercourse. This is a substance that once applied to the vagina, turns into a mixture of estrogen and testosterone. We know from prior research that the vestibule area is rich in testosterone receptors, so it makes sense that DHEA cream applied vaginally would be able to help vulvodynia patients. However, we do not know the ratio of the breakdown of estrogen versus testosterone from the DHEA substance.

Testosterone applied to the vagina has been shown to improve symptoms in patients with other vulvar conditions, such as lichen sclerosus. Lichen sclerosus is a chronic skin condition that primarily affects the genital area, but it can also affect other areas of the body. It is characterized by white, thickened patches of skin that may be itchy, sore, or painful.

Although topical DHEA was FDA approved for use in women with painful intercourse in 2016, topical testosterone combined with estrogen is not FDA approved for use in women, which means it is investigational. However, it is becoming more common as a treatment option for patients with vulvodynia, and its safety and effectiveness in women has been demonstrated in other studies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients with vulvodynia who present with pain (with vaginal penetration) rating score of 4 or greater

Exclusion Criteria:

* Active vaginal infection
* Pregnancy
* Breast-feeding
* Taking anti-androgenic medication (finasteride, dutasteride)
* Using any other topical hormones to the vulva or vagina

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Typical pain with vaginal penetration within last 2 weeks | at 12 weeks post-treatment
  Typical pain with vaginal penetration within last 2 weeks using numeric rating scale

SECONDARY OUTCOMES:
Typical pain with vaginal penetration within last 2 weeks | at 6 weeks post-treatment
  Typical pain with vaginal penetration within last 2 weeks using numeric rating scale
Sexual function | at 6 weeks and 12 weeks post-treatment
  sexual function as measured by Female Sexual Function Index
Most intense pain with vaginal penetration within last 2 weeks | at 6 weeks and 12 weeks post-treatment
  Most intense pain with vaginal penetration within last 2 weeks using numeric rating scale

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Urogynecology Associates, Cincinnati, Ohio
  - TriHealth, Cincinnati, Ohio